CLINICAL TRIAL: NCT05217212
Title: Do Markers of Systemic Inflammatory Response and Tumor Metabolism Indicate Radioresistance in Head and Neck Cancer?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Universität Luzern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00317
Record Dates: First submitted 2021-12-30; First posted 2022-02-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiochemotherapy — Primary radiotherapy of the primary tumor and nodal basin with curative intent with or without concomitant chemotherapy with cisplatin, carboplatin, or cetuximab weekly.

SUMMARY:
The aim of the study is to prospectively evaluate whether markers of a patient's systemic inflammatory response in addition to FDG-PET/CT metabolic parameters of the primary tumor or of nodal metastases can predict radioresistance and survival before primary radiochemotherapy in advanced head and neck cancer patients.

DETAILED DESCRIPTION:
This study prospectively investigates pretherapeutic markers of systemic inflammatory response (including neutrophil-to-lymphocyte ratio, platelet-to-lymphocyte ratio, lymphocyte-to-monocyte ratio, systemic inflammation response index, and systemic immune-inflammation) and FDG-PET/CT-derived metabolic parameters of tumor and nodal metastases (including maximum standardized uptake value, metabolic tumor volume, and total lesion glycolysis) and their potential prognostic value in head and neck cancer patients prior to primary radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histopathologic diagnosis of squamous cell carcinoma of the head and neck
* primary radio(chemo)therapy with curative intent
* available pretherapeutic FDG-PET/CT imaging
* available pretherapeutic differential blood analysis

Exclusion Criteria:

* other tumor entities of the head and neck including cutaneous squamous cell carcinoma
* primary surgical treatment
* ongoing infections or other inflammatory diseases at the time of diagnosis
* patients not completing a course of irradiation with at least 66 Gray locally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing primary radio(chemo)therapy for oral, oropharyngeal, epipharyngeal, hypopharyngeal or laryngeal squamous cell carcinoma at Cantonal Hospital Lucerne, Switzerland
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survival | Prospective analysis of various measures of survival up to 5 years after completion of the therapy. Events such as tumor recurrence or death will be recorded continually.
  Overall survival, disease-specific survival, local and regional recurrence-free survival, and distant metastasis-free survival

OTHER OUTCOMES:
Correlation Analysis | At diagnosis
  Analysis of a correlation of pretherapeutic systemic inflammatory markers in differential blood analysis including neutrophil-to-lympocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), lym-phocyte-to-monocyte ratio (LMR), systemic immune-inflammation index (SII), and systemic in-flammation response index (SIRI) and FDG-PET/CT-derived parameters of tumor metabolism such as maximum standardized uptake value (SUVmax), total lesion glycolysis (TLG), and metabolic tumor volume (MTV) of the primary tumor and lymph node metastases.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology - Head and Neck Surgery, Cantonal Hospital Lucerne, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No